CLINICAL TRIAL: NCT02406703
Title: Can the Choice of the Local Anesthetic Have an Impact on Ambulatory Surgery Perioperative Costs? Chloroprocaine for Popliteal Block in Outpatient Foot Surgery
Brief Title: The Impact of Chloroprocaine 3% for Ambulatory Foot Surgery on Perioperative Process Costs
Status: Completed | Type: Observational
Sponsor: Ospedale Regionale Bellinzona e Valli (Other)
Responsible Party: Principal Investigator, Andrea Saporito, MD, Ospedale Regionale Bellinzona e Valli
Other Study IDs: BLV07
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Impact of Anesthetic Choice on Costs
Keywords: local anesthesia; regional anesthetic
MeSH Terms: interventions — chloroprocaine; Mepivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chloroprocaine: Patient undergoing popliteal block with chloroprocaine
  Interventions: Drug: Chloroprocaine
- Mepivacaine: Patient undergoing popliteal block with mepivacaine
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Drug: Chloroprocaine
  Groups: Chloroprocaine
Drug: Mepivacaine
  Groups: Mepivacaine

SUMMARY:
Background and Objectives Short acting regional anesthetics have already been successfully employed for peripheral nerve blocks in an ambulatory surgery setting. However, the impact on direct and indirect perioperative costs comparing two different short-acting local anesthetics has not been performed, yet.

Methods In an observational study including 50 patients per group, patient undergoing popliteal block with chloroprocaine 3% or mepivacaine 1.5% for ambulatory minor foot surgery were compared. The primary outcome was the saving of both direct and indirect perioperative costs. Secondary outcomes were block success, onset time and block duration, patient satisfaction and unplanned outpatient visits or readmissions after discharge.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III scheduled for elective, unilateral, ambulant minor foot surgery (percutaneous hallux valgus correction, osteotomies, tenotomies, mallet and hammer toes correction, screws and/or plaques removal)

Exclusion Criteria:

* known allergy to drugs used in the study;
* coagulopathies, known neuropathy;
* pregnancy;
* chronic pain;
* drug or alcohol abuse;
* psychiatric disease or lack of competence affecting compliance and evidence of ongoing sepsis or local skin / subcutaneous tissues infections in the popliteal fossa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-III scheduled for elective, unilateral, ambulant minor foot surgery (percutaneous hallux valgus correction, osteotomies, tenotomies, mallet and hammer toes correction, screws and/or plaques removal)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cost minimization analysis | 6 months